CLINICAL TRIAL: NCT05652374
Title: Gag Therapy for Recurrent Urinary Tract Infection Assessing Comparability to International Nitrofurantoin Gold Standard Study
Acronym: GT RACING
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: IBSA Institut Biochimique SA (Industry); Goodlife Pharma B.V. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 111802; NL76892.091.21 (Other: algemeen beoordelings- en registratie)
Record Dates: First submitted 2022-11-23; First posted 2022-12-15 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-07

CONDITIONS: Recurrent Urinary Tract Infection
Keywords: GAG therapy; Prophylactic antibiotics
MeSH Terms: conditions — Urinary Tract Infections | interventions — Nitrofurantoin

STUDY DESIGN:
Intervention Model Description: Cross-over randomized controlled trial. Study is set-up as non-inferiority, parallel group trial, with a 1:1 randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Other): Ialuril therapy for 6 months followed by nitrofuranoïne (or trimethoprim) prophylactic therapy for 6 months. In between therapies there is a 4 week wash-out period.
  Interventions: Device: Ialuril 50ml Prefill; Drug: Nitrofurantoin
- Group B (Other): Nitrofuranoïne (or trimethoprim) prophylactic therapy for 6 months followed by Ialuril therapy for 6 months. In between therapies there is a 4 week wash-out period.
  Interventions: Device: Ialuril 50ml Prefill; Drug: Nitrofurantoin

INTERVENTIONS:
Device: Ialuril 50ml Prefill — 50ml of sterile Ialuril (HA 1.6% CS 2%) bladder instillations weekly for 6 weeks, followed by monthly maintenance therapy for 6 months
  Other Names: HA-CS
Drug: Nitrofurantoin — nitrofurantoin 100mg daily (1dd100mg or 2dd50mg) for 6 months. ( In case of resistance/intolerance/allergy for nitrofurantoin alternatively trimethoprim 100mg daily)

SUMMARY:
The GT RACING is a study comparing the efficacy of HA-CS bladder installations with prophylactic antibiotics in the prevention of recurrent urinary tract infections (rUTI).

DETAILED DESCRIPTION:
The main objective of the study is to compare efficacy between hyaluronic acid - chondroitin sulphate (HA-CS) treatment and gold standard treatment (AB prophylaxis). Study is set-up as non-inferiority, parallel group cross-over RCT, with a 1:1 randomization.

Study population: Female (>18rs) with at least 3 symptomatic urinary tract infections (UTI's) in the previous year with no adequate curable therapeutic options.

Intervention: 50ml of sterile Ialuril (HA 1.6% CS 2%) weekly for 6 weeks, followed by monthly maintenance therapy for 6 months.

Control : oral nitrofurantoin 100mg daily (1dd100mg or 2dd50mg) for 6 months. In case of resistance/intolerance/allergy for nitrofurantoin alternatively trimethoprim 100mg daily will be given.

All patients recieve both treatments (ialuril and nitrofurantoin) consecutively, for 6 months each. The order of the therapies is determined by randomisation. Between therapies there is a 4 weeks 'wash-out' period. A total of 100 patients will be included.

During the study patients will fill-out questionnaires regarding symptoms, quality of life and use of healthcare. Furthermore urine will be collected at set timepoints.

Main study parameters/endpoints: The main study parameter is the number of UTI per patient-year. Secondary parameters are time to rUTI (wks.), outcome on the global responce assessment (GRA) scale, pattern of antibiotic resistance, outcome on the patient reported outcome questionnaire, cost effectiveness and Quality-of-life.

ELIGIBILITY:
Inclusion Criteria:

1. Adult female patients (>18 years) who had at least 3 symptomatic UTI's in the previous year with no adequate curable therapeutic options (e.g. bladder stones)
2. At least one UTI's must be confirmed with a positive culture and antibiogram, further UTI's must be confirmed with a urine sediment with positive nitrite or a positive culture.

Exclusion Criteria:

1. Male
2. < 18 years
3. Pregnant
4. Already on GAG therapy
5. Already on prophylactic antibiotics
6. Started or stopped cranberry/d-mannose therapy or vaginal estrogenic creme in the last two months
7. Had Gentamicin or other antibiotic instillations in the previous 2 months
8. Allergic to >3 regular used antibiotics in Dutch guidelines (ed. Nitrofurantoin, trimethoprim, Fosfomycin)
9. A urinary fistula
10. Urinary stones
11. Urogenital cancer
12. Bladder Pain Syndrome - Interstitial Cystitis
13. Chronic pelvic pain
14. Had a STD untreated or treated in the previous 2 months
15. A urinary diversion
16. An Indwelling catheter
17. A suprapubic catheter
18. Performing >1/day self-catheterization
19. A residue after voiding (PVR) of >200ml
20. Unable (also legal) to give informed consent
21. Recurrent urosepsis
22. Multiresistant bacteria in previous urine cultures
23. Contra-indications and interactions for Nitrofurantoin: severe kidney disfunction (GFR < 30), lung- or liver problems or neuropathy after previous use of nitrofurantoin, acute porphyria, known G6PD deficiency, use of magnesium trisilicate.
24. Contra-indications and interactions for trimethoprim: severe kidney or liver dysfunction, blood count abnormality, use of vitamin K antagonists, use of folic acid antagonists, use of ace inhibitors
25. Severe lung/respiratory disfunction (reduced lung capacity, lung cancer, fibrosis, COPD)
26. Does not tolerate catheterization

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-10-20 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Number of urinary tract infections | 13 months
  Number of urinary tract infections per patient-year

SECONDARY OUTCOMES:
Time to first urinary tract infection | 13 months
  Time to first urinary tract infection
Global Assessment of Improvement | 7 weeks, 3 months, 6 months after start of each therapy
  Changes on Global Assessment of Improvement, Likert scale: -3 (worst) to +3(best)
Antibiotics resistance | Baseline, 6 months after start of each therapy
  Difference in acquired AB resistance (increase in resistance to different antibiotic treatments) between both patients groups
Cost-effectiveness: medical consumption questionnaire | Baseline, 6 months after start of each therapy
  Difference in cost-effectiveness between the 2 therapies. This is assessed with the 'medical consumption questionnaire'
Cost-effectiveness: productivity cost questionnaire | Baseline, 6 months after start of each therapy
  Difference in cost-effectiveness between the 2 therapies. This is assessed with the 'productivity cost questionnaire'
Therapy specific patient reported outcomes (symptoms & bother) | baseline, 7 weeks, 3 months, 6 months after start of each therapy
  Differences in therapy specific patient reported outcomes between both patient groups (measured in Therapy Specific Patient Reported Outcome (PRO) Questionnaire on Symptom & Bother rUTI & GAG therapy)
General quality of life questionnaire (mobility, self-care, daily activities, pain/discomfort, anxiety/depression) | baseline, 7 weeks, 3 months, 6 months after start of each therapy
  Is there a difference in the Quality-of-life between the 2 therapies during follow-up using ED-5D 5L questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Dick Janssen, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (3):
- Netherlands (3):
  - Radboudumc, Nijmegen, Gelderland
  - Rijnstate ziekenhuis, Arnhem
  - Canisius wilhelmina ziekenhuis, Nijmegen

IPD SHARING:
Plan to Share IPD: No
only anonymous patient data will be shared